CLINICAL TRIAL: NCT03858803
Title: Improving the Reproductive Health of Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Botswana Study
Record Dates: First submitted 2019-02-21; First posted 2019-03-01 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Reproductive Health
Keywords: HIV; STI; Unplanned pregnancy; Reproductive health of families; Adolescents
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Random assignment to one of three experimental arms:
  Arm 1: Parents complete intervention immediately, adolescents complete intervention 6 month later Arm 2: Both parents and adolescents participate in intervention simultaneously Arm 3: Comparison condition in which both parents and adolescents are offered their respective interventions after the final assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FM2 first, LAST delayed (Active Comparator): Parent intervention, Families Matter 2 (FM2), immediate, adolescent intervention, Living as a Safer Teen (LAST), delayed six months
  Interventions: Behavioral: Families Matter 2; Behavioral: Living as a Safer Teen
- FM2 and LAST simultaneous (Active Comparator): Parents participate in Families Matter 2 (FM2) and adolescents in Living as a Safer Teen (LAST) intervention immediately following the baseline assessment.
  Interventions: Behavioral: Families Matter 2; Behavioral: Living as a Safer Teen
- Comparison arm (Active Comparator): Comparison arm in which both parents and adolescents will be offered their respective interventions following the final assessment. Following the final assessment parents will be offered the Families Matter (FM2) intervention and youth the Living as a Safer Teen (LAST) intervention as an ethically justified service.
  Interventions: Behavioral: Families Matter 2; Behavioral: Living as a Safer Teen

INTERVENTIONS:
Behavioral: Families Matter 2 — Parents training in communication, youth sexual development, parental monitoring, parental use of positive reinforcement, risks facing adolescents and their management.
  Other Names: FM2
Behavioral: Living as a Safer Teen — Prevention intervention for adolescents 13-18 that provides information, motivation, and behavioral skills to prevent STIs, HIV, and unplanned pregnancy.
  Other Names: LAST

SUMMARY:
This research will assess the effectiveness of a parent- and an adolescent- intervention in lowering risk of STIs, HIV, and unintended pregnancies among Batswana youth.

DETAILED DESCRIPTION:
Youth in Botswana face extraordinary challenges as they transition through adolescence. High rates of teen pregnancy force girls to drop out of school after which few resume their education. Sexually transmitted infections (STIs) are prevalent and the country has the 3rd highest Human Immunodeficiency Virus (HIV) prevalence in the world, with incidence increasing rapidly among adolescents 15-19, peaking at 40.2% HIV seroprevalence at ages 30-34. Traditional methods for sex education through village initiation schools are no longer available and parents are not comfortable with discussions addressing reproductive health within the family. As a result, adolescents have no conduit to educate them about healthy sexual development. This study will recruit 456 families, ½ with a male and ½ with a female adolescent. Families will be randomized to one of three intervention arms. Parents will participate in Families Matter 2! (FM2) and adolescents in Living as a Safer Teen (LAST), both evidence-based interventions that were adapted and pilot tested in Botswana during an earlier R34 award. In Arm 1, the parent will participate in FM2 immediately and the youth will participate in LAST six months later. In Arm 2, both the parent and youth will participant in their respective interventions simultaneously. In Arm 3, the comparison condition, participants will be offered the interventions immediately after the final assessment. Each adolescent and parent will complete assessments in English or Setswana at baseline, post-intervention, and 6- and 12-month follow-ups. Results from a pilot trial of the adapted interventions suggest that these interventions may result in improved family communications, child management skills, knowledge of sexual development, more favorable attitudes toward contraception, less tolerance for intergenerational transactional sex, greater rejection of gender violence, and lower rates of sexual risk behavior by both parents and adolescents. It is further anticipated that youths who are abstinent upon entering the intervention will delay sexual debut to a greater extent than youth in the comparison arm. This proposed study addresses the highest priority in Botswana's current national strategic plan: preventing early pregnancy, STIs and HIV in adolescents. If the proposed randomized controlled trial (RCT) provides strong evidence of effectiveness, the investigators will work with the Ministries of Education, Health, Youth & Culture and the Office of the President to disseminate the intervention throughout Botswana.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent 13-18 in or near Gaborone Botswana and parent/guardian

Exclusion Criteria:

* None

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 945 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet S St. Lawrence, Ph.D., Principal Investigator — Portland State University; Esther S Seloilwe, Ph.D., Study Director — University of Botswana
Locations (1):
- Janet S. St. Lawrence, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be made available upon study completion.

RESULTS

PARTICIPANT FLOW:
Groups:
- FM2 First, LAST Delayed - Youth; FM2 First, LAST Delayed - Parents: Parent intervention, Families Matter 2 (FM2), immediate, adolescent intervention, Living as a Safer Teen (LAST), delayed six months
  Families Matter 2: Parents training in communication, youth sexual development, parental monitoring, parental use of positive reinforcement, risks facing adolescents and their management.
  Living as a Safer Teen: Prevention intervention for adolescents 13-18 that provides information, motivation, and behavioral skills to prevent STIs, HIV, and unplanned pregnancy.
- FM2 and LAST Simultaneous - Youth; FM2 and LAST Simultaneous - Parents: Parents participate in Families Matter 2 (FM2) and adolescents in Living as a Safer Teen (LAST) intervention immediately following the baseline assessment.
  Families Matter 2: Parents training in communication, youth sexual development, parental monitoring, parental use of positive reinforcement, risks facing adolescents and their management.
  Living as a Safer Teen: Prevention intervention for adolescents 13-18 that provides information, motivation, and behavioral skills to prevent STIs, HIV, and unplanned pregnancy.
- Comparison Arm - Youth; Comparison Arm - Parents: Comparison arm in which both parents and adolescents will be offered their respective interventions following the final assessment. Following the final assessment parents will be offered the Families Matter (FM2) intervention and youth the Living as a Safer Teen (LAST) intervention as an ethically justified service.
  Families Matter 2: Parents training in communication, youth sexual development, parental monitoring, parental use of positive reinforcement, risks facing adolescents and their management.
  Living as a Safer Teen: Prevention intervention for adolescents 13-18 that provides information, motivation, and behavioral skills to prevent STIs, HIV, and unplanned pregnancy.
Period: Overall Study
Arm/Group | FM2 First, LAST Delayed - Youth | FM2 First, LAST Delayed - Parents | FM2 and LAST Simultaneous - Youth | FM2 and LAST Simultaneous - Parents | Comparison Arm - Youth | Comparison Arm - Parents
Started | 161 | 161 | 158 | 160 | 153 | 152
Post | 161 | 161 | 158 | 160 | 153 | 152
Completed | 148 | 151 | 153 | 155 | 149 | 149
Not Completed | 13 | 10 | 5 | 5 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Comparison Arm - Parents: Comparison arm in which both parents and adolescents will be offered their respective interventions following the final assessment. Following the final assessment parents will be offered the Families Matter (FM2) intervention and youth the Living as a Safer Teen (LAST) intervention as an ethically justified service.
- Total: Total of all reporting groups
Arm/Group | FM2 First, LAST Delayed - Youth | FM2 and LAST Simultaneous - Youth | Comparison Arm - Youth | FM2 First, LAST Delayed - Parents | FM2 and LAST Simultaneous - Parents | Comparison Arm - Parents | Total
Number analyzed (Participants) | 161 | 158 | 153 | 161 | 160 | 152 | 945
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 161 | 158 | 153 | 0 | 3 | 2 | 477
  Between 18 and 65 years | 0 | 0 | 0 | 154 | 153 | 143 | 450
  >=65 years | 0 | 0 | 0 | 7 | 4 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (1.7) | 15.26 (1.5) | 15.00 (1.7) | 41.95 (9.12) | 38.56 (9.34) | 41.03 (9.79) | 27.83 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 86 | 84 | 142 | 143 | 139 | 689
  Male | 66 | 72 | 69 | 19 | 17 | 13 | 256
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 161 | 158 | 153 | 161 | 160 | 152 | 945
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Botswana | 161 | 158 | 153 | 161 | 160 | 152 | 945
Parental Monitoring [Mean (Standard Deviation); unit: units on a scale] — Total scale score range 0-16, No subscales, Higher scores reflect report of greater parental monitoring
  units on a scale | 9.51 (3.75) | 10.03 (4.25) | 9.62 (4.24) | 8.35 (4.22) | 8.38 (4.48) | 8.20 (4.63) | 9.02 (.72)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Frequency of Unprotected Intercourse (Youth)
Description: Self-reported frequency of unprotected intercourse occasions in past 3 months.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: number of occassions
Arm/Group | FM2 First, LAST Delayed | FM2 and LAST Simultaneous | Comparison Arm
Number analyzed (Participants) | 148 | 153 | 149
number of occassions | 1.42 (3.09) | 1.16 (1.78) | 1.38 (2.93)
Statistical Analysis 1: Comparison: FM2 First, LAST Delayed vs FM2 and LAST Simultaneous vs Comparison Arm; Test type: Superiority; p < .05, MANOVA

2. Primary Outcome: Changes in Reproductive Health Knowledge Test Scores (Youth)
Description: Measure of knowledge about prevention of STIs, HIV, and pregnancy. Total score range 0-26. No subscales. Higher scores reflect more accurate knowledge.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FM2 First, LAST Delayed | FM2 and LAST Simultaneous | Comparison Arm
Number analyzed (Participants) | 148 | 153 | 149
score on a scale | 12.79 (6.32) | 14.66 (6.90) | 11.37 (5.99)
Statistical Analysis 1: Comparison: FM2 First, LAST Delayed vs FM2 and LAST Simultaneous vs Comparison Arm; Test type: Superiority; p < .05, MANOVA

3. Primary Outcome: Changes in Condom Barriers Scale(Youth)
Description: Total score range 0 - 140; Higher scores reflect greater perceived barriers to condom use. No subscales
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FM2 First, LAST Delayed | FM2 and LAST Simultaneous | Comparison Arm
Number analyzed (Participants) | 148 | 153 | 149
score on a scale | 63.67 (20.08) | 57.73 (22.30) | 66.37 (19.12)
Statistical Analysis 1: Comparison: FM2 First, LAST Delayed vs FM2 and LAST Simultaneous vs Comparison Arm; Test type: Superiority; p < .05, MANOVA

4. Primary Outcome: Change in Attitudes Toward Transactional Sex Scale (Youth)
Description: Total score range 0 - 120, No subscales, Higher scores reflect more acceptance of transactional sex
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FM2 First, LAST Delayed | FM2 and LAST Simultaneous | Comparison Arm
Number analyzed (Participants) | 148 | 153 | 149
score on a scale | 19.67 (12.93) | 20.44 (13.49) | 23.18 (14.70)
Statistical Analysis 1: Comparison: FM2 First, LAST Delayed vs FM2 and LAST Simultaneous vs Comparison Arm; Test type: Superiority; p < .05, MANOVA

5. Primary Outcome: Change in Number of Sex Partners (Youth)
Description: Change in self-reported numbers of sex partners in past two months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of sex partners
Arm/Group | FM2 First, LAST Delayed | FM2 and LAST Simultaneous | Comparison Arm
Number analyzed (Participants) | 148 | 153 | 149
number of sex partners | 0.91 (0.80) | 1.12 (2.09) | 2.14 (3.59)
Statistical Analysis 1: Comparison: FM2 First, LAST Delayed vs FM2 and LAST Simultaneous vs Comparison Arm; Test type: Superiority; p < .05, MANOVA

6. Primary Outcome: Changes on Family Communication Scale (Youth)
Description: Total scale range 0-52, No subscales, Higher scores reflect more frequent communication between parent and child frequency
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FM2 First, LAST Delayed | FM2 and LAST Simultaneous | Comparison Arm
Number analyzed (Participants) | 148 | 153 | 149
score on a scale | 23.89 (14.58) | 24.33 (14.53) | 20.73 (13.82)
Statistical Analysis 1: Comparison: FM2 First, LAST Delayed vs FM2 and LAST Simultaneous vs Comparison Arm; Test type: Superiority; p < .05, MANOVA

7. Primary Outcome: Changes in Scores on the Condom Attitudes Scale (Youth)
Description: Total scale score range 0-144, No subscales, Higher scores reflect more positive attitudes toward condom use
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FM2 First, LAST Delayed | FM2 and LAST Simultaneous | Comparison Arm
Number analyzed (Participants) | 148 | 153 | 149
score on a scale | 94.40 (26.50) | 96.65 (31.00) | 92.09 (26.85)
Statistical Analysis 1: Comparison: FM2 First, LAST Delayed vs FM2 and LAST Simultaneous vs Comparison Arm; Test type: Superiority; p < .05, MANOVA

8. Primary Outcome: Changes in Scores on Self Efficacy Beliefs Scale (Youth)
Description: Total scale score range 0-160, No subscales, Higher scores reflect endorsement of greater self efficacy beliefs
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FM2 First, LAST Delayed | FM2 and LAST Simultaneous | Comparison Arm
Number analyzed (Participants) | 148 | 153 | 149
score on a scale | 58.99 (47.29) | 71.82 (52.68) | 67.83 (52.05)
Statistical Analysis 1: Comparison: FM2 First, LAST Delayed vs FM2 and LAST Simultaneous vs Comparison Arm; Test type: Superiority; p < .05, MANOVA

9. Primary Outcome: Changes on Parental Responsiveness Scale (Youth)
Description: Total scale score range 0-11, No subscales, Higher scores reflect reports of greater parental responsiveness
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FM2 First, LAST Delayed | FM2 and LAST Simultaneous | Comparison Arm
Number analyzed (Participants) | 148 | 153 | 149
score on a scale | 6.06 (3.72) | 6.41 (3.59) | 5.23 (3.70)
Statistical Analysis 1: Comparison: FM2 First, LAST Delayed vs FM2 and LAST Simultaneous vs Comparison Arm; Test type: Superiority; p < .05, MANOVA

10. Primary Outcome: Changes in Parent Use of Positive Reinforcement Scale (Youth)
Description: Total score range 0-12, No Subscales, Higher score reflect reports of more frequent use of positive reinforcement by parents
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FM2 First, LAST Delayed | FM2 and LAST Simultaneous | Comparison Arm
Number analyzed (Participants) | 148 | 153 | 149
score on a scale | 5.95 (3.11) | 5.92 (3.23) | 5.78 (3.26)
Statistical Analysis 1: Comparison: FM2 First, LAST Delayed vs FM2 and LAST Simultaneous vs Comparison Arm; Test type: Superiority; p < .05, MANOVA

11. Primary Outcome: Changes in Parental Monitoring Scale (Youth)
Description: Total scale score range 0-16, No subscales, Higher scores reflect report of greater parental monitoring
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FM2 First, LAST Delayed | FM2 and LAST Simultaneous | Comparison Arm
Number analyzed (Participants) | 148 | 153 | 149
score on a scale | 9.67 (3.92) | 9.82 (4.43) | 10.03 (3.93)
Statistical Analysis 1: Comparison: FM2 First, LAST Delayed vs FM2 and LAST Simultaneous vs Comparison Arm; Test type: Superiority; p < .05, MANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- FM2 First, LAST Delayed - Parent: Parent intervention, Families Matter 2 (FM2), immediate, adolescent intervention, Living as a Safer Teen (LAST), delayed six months
  Families Matter 2: Parents training in communication, youth sexual development, parental monitoring, parental use of positive reinforcement, risks facing adolescents and their management.
  Living as a Safer Teen: Prevention intervention for adolescents 13-18 that provides information, motivation, and behavioral skills to prevent STIs, HIV, and unplanned pregnancy.
- FM2 and LAST Simultaneous - Parent: Parents participate in Families Matter 2 (FM2) and adolescents in Living as a Safer Teen (LAST) intervention immediately following the baseline assessment.
  Families Matter 2: Parents training in communication, youth sexual development, parental monitoring, parental use of positive reinforcement, risks facing adolescents and their management.
  Living as a Safer Teen: Prevention intervention for adolescents 13-18 that provides information, motivation, and behavioral skills to prevent STIs, HIV, and unplanned pregnancy.
- Comparison Arm - Parent: Comparison arm in which both parents and adolescents will be offered their respective interventions following the final assessment. Following the final assessment parents will be offered the Families Matter (FM2) intervention and youth the Living as a Safer Teen (LAST) intervention as an ethically justified service.
  Families Matter 2: Parents training in communication, youth sexual development, parental monitoring, parental use of positive reinforcement, risks facing adolescents and their management.
  Living as a Safer Teen: Prevention intervention for adolescents 13-18 that provides information, motivation, and behavioral skills to prevent STIs, HIV, and unplanned pregnancy.
Arm/Group | FM2 First, LAST Delayed - Youth | FM2 and LAST Simultaneous - Youth | Comparison Arm - Youth | FM2 First, LAST Delayed - Parent | FM2 and LAST Simultaneous - Parent | Comparison Arm - Parent
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/158 | 0/153 | 0/161 | 0/160 | 0/152
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/158 | 0/153 | 0/161 | 0/160 | 0/152
Other Adverse Events (participants affected / at risk) | 0/161 | 0/158 | 0/153 | 0/161 | 0/160 | 0/152

LIMITATIONS AND CAVEATS:
One year follow-up for intervention outcomes was planned; however, the COVID pandemic and associated restrictions interrupted data collection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT03858803/Prot_SAP_000.pdf